CLINICAL TRIAL: NCT04259918
Title: Effect of Alveolar Recruitment Maneuver on Postoperative Pain After Bariatric Surgery
Brief Title: Effect of Alveolar Recruitment Maneuver on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gil2019-1
Record Dates: First submitted 2020-01-20; First posted 2020-02-07 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: enrolled groups ares only selected and applied in the operating room and participants, care giver and outcomes accessor could not know the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): no applying alveolar recuritment maneuver
  Interventions: Procedure: Alveolar recruitment maneuver
- Low ARM (Active Comparator): Applying 30 cmH2O of alveolar recruitment maneuver 5 times every 5sec
  Interventions: Procedure: Alveolar recruitment maneuver
- High ARM (Active Comparator): Applying 60 cmH2O of alveolar recruitment maneuver 5 times every 5sec
  Interventions: Procedure: Alveolar recruitment maneuver

INTERVENTIONS:
Procedure: Alveolar recruitment maneuver — Applying 30 or 60 cmH2O of alveolar recruitment maneuver 5 times every 5 min at the end of bariatric surgery
  Other Names: Low pressure alveolar recruitment maneuver; High pressure alveolar recruitment maneuver

SUMMARY:
Control group: no additional procedure Low ARM group : recruitment maneuver of 30cmH2O High ARM group: recruitment maneuver of 60cmH2O

DETAILED DESCRIPTION:
After random assignment of group, Control group: no additional procedure apply, Low ARM group : after surgical trocha out after bariatric surgery, applying 30cmH2O recruitment maneuver 5 times every 5 seconds, High ARM group: after surgical trocha out after bariatric surgery, applying 60cmH2O recruitment maneuver 5 times every 5 seconds

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled for elective bariatric surgery

Exclusion Criteria:

* uncontrolled cardio-vascular disease, active pulmonary disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-25 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale for postoperative pain | up to postoperative 24 hour
  score (0 no pain-10 severe pain)
Quality of recovery (QoR40) for Postoperative comfort | up to postoperative 24 hour
  score 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery)